CLINICAL TRIAL: NCT06567964
Title: Comparative Efficacy of Ultrasound-guided Erector Spinae Plane Block Versus Wound Infiltration for Postoperative Analgesia in Instrumented Lumbar Spinal Surgeries
Brief Title: Ultrasound-guided ESP Block vs. Wound Infiltration in Lumbar Surgery: A Comparative Analysis (ESP:Erector Spinae Plane)
Acronym: ESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YÜCEL YÜCE, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SaglikBilimleriU-KLKSH-Anes-02
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Spine Instability; Lumbar Spine Degeneration
Keywords: Erector Spinae Plane Block; Wound Infiltration; Postoperative Analgesia; Lumbar Spinal Surgery; Ultrasound-Guided Anesthesia; Postoperative Pain; Visual Analog Scale (VAS); Enhanced Recovery After Surgery (ERAS)
MeSH Terms: conditions — Spinal Stenosis; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants
  Eligible participants were adults aged 18-70 years who were scheduled for elective lumbar spinal surgery with instrumentation. The inclusion criteria were as follows:
  * Elective lumbar spine surgery involving instrumentation
  * ASA physical status I-III
  * Ability to provide informed consent
  The exclusion criteria were as follows:
  * Known allergies to local anesthetics
  * Coagulopathy or anticoagulant therapy
  * Infection at the injection site
  * Preexisting neurological disorders affecting sensory perception
  * Pregnancy
  * Inability to understand the visual analog scale (VAS) for pain assessment The participants were randomly allocated into one of two groups: the ESPB group (Group E) or the WI group (Group W).
Who Masked: Participant, Outcomes Assessor
Masking Description: Randomization and Blinding A computer-generated random number sequence was used for randomization. Allocation was concealed via sealed, opaque envelopes, which were opened just before the intervention. Both the patients and the outcome assessors were blinded to the group assignments. The anesthesiologist who administered the block was aware of the group allocation but did not participate in the postoperative assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Group E) (Active Comparator): ESPB was administered preoperatively under ultrasound guidance via a high-frequency linear probe (Sonosite M-Turbo, Fujifilm Sonosite Inc., USA) (Figure 1). The procedure was as follows:
  1. Patient Positioning: The patient was positioned in the lateral decubitus position, with the side to be blocked uppermost.
  2. Ultrasound Setup: A high-frequency linear ultrasound probe was placed in a parasagittal orientation over the transverse process of the lumbar vertebra at the level of surgery.
  3. Needle Insertion: After skin disinfection with chlorhexidine, a 22-gauge, 100-mm needle (Stimuplex A, B. Braun Melsungen AG, Germany) was inserted in-plane to the ultrasound probe. The needle was advanced until the tip contacted the transverse process.
  4. Injection: Following negative aspiration to ensure no vascular puncture, 20 mL of 0.5% bupivacaine was injected incrementally, with real-time ultrasound visualization to confirm the correct spread of the anesthetic solution.
  Interventions: Procedure: Erector Spinae Plane Block(ESPB)
- Wound infiltration (Group WI) (Active Comparator): Wound infiltration was performed by the surgeon at the end of the surgery via the following procedure:
  1. Preparation: After hemostasis was achieved and before skin closure, 20 mL of 0.5% bupivacaine was prepared in a sterile syringe.
  2. For infiltration, the anesthetic mixture was infiltrated into multiple layers of the surgical wound. This included the subcutaneous tissue and muscle layers, ensuring the even distribution of the anesthetic solution to cover the entire surgical area.
  Interventions: Procedure: Wound infiltration

INTERVENTIONS:
Procedure: Erector Spinae Plane Block(ESPB) — ESPB was administered preoperatively under ultrasound guidance via a high-frequency linear probe (Sonosite M-Turbo, Fujifilm Sonosite Inc., USA) (Figure 1). The procedure was as follows:
  1. Patient Positioning: The patient was positioned in the lateral decubitus position, with the side to be blocked uppermost.
  2. Ultrasound Setup: A high-frequency linear ultrasound probe was placed in a parasagittal orientation over the transverse process of the lumbar vertebra at the level of surgery.
  3. Needle Insertion: After skin disinfection with chlorhexidine, a 22-gauge, 100-mm needle (Stimuplex A, B. Braun Melsungen AG, Germany) was inserted in-plane to the ultrasound probe. The needle was advanced until the tip contacted the transverse process.
  4. Injection: Following negative aspiration to ensure no vascular puncture, 20 mL of 0.5% bupivacaine was injected incrementally, with real-time ultrasound visualization to confirm the correct spread of the anesthetic solution.
  Arms: Erector Spinae Plane Block (Group E)
Procedure: Wound infiltration — Wound infiltration was performed by the surgeon at the end of the surgery via the following procedure:
  1. Preparation: After hemostasis was achieved and before skin closure, 20 mL of 0.5% bupivacaine was prepared in a sterile syringe.
  2. For infiltration, the anesthetic mixture was infiltrated into multiple layers of the surgical wound. This included the subcutaneous tissue and muscle layers, ensuring the even distribution of the anesthetic solution to cover the entire surgical area.
  Arms: Wound infiltration (Group WI)

SUMMARY:
This study aimed to compare the efficacy of ultrasound-guided erector spinae plane block (ESPB) with that of wound infiltration (WI) for postoperative analgesia in lumbar spinal surgeries involving instrumentation.

DETAILED DESCRIPTION:
In this randomized controlled trial, 80 patients were divided into two groups: ESPB (n=40) and WI (n=40). Postoperative pain intensity was assessed using the Visual Analog Scale (VAS) at multiple time points within 24 hours. Additionally, opioid consumption, time to first rescue analgesia, incidence of postoperative nausea and vomiting (PONV), and patient satisfaction were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Elective lumbar spine surgery involving instrumentation
* ASA physical status I-III
* Ability to provide informed consent

Exclusion Criteria:

* Known allergies to local anesthetics
* Coagulopathy or anticoagulant therapy
* Infection at the injection site
* Preexisting neurological disorders affecting sensory perception
* Pregnancy
* Inability to understand the visual analog scale (VAS) for pain assessment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity | 1., 6., 12., 24., and 48. hours postoperatively
  The pain intensity was assessed via the visual analog scale (VAS).The VAS is a 10 cm scale ranging from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Total Opioid Consumption | In the first 48 hours postoperatively
  Recorded as morphine equivalents
Time to first request for rescue analgesia | Noted in hours in the first 48 hours postoperatively
  Noted in hours postoperatively
Incidence of Side Effects | Recorded as binary outcomes (present/absent) in the first 48 hours postoperatively
  Including nausea, vomiting, pruritus, and urinary retention,
Patient Satisfaction with Pain Management | At 48 hours postoperatively
  Patient satisfaction was assessed via a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Yücel Yüce, MD,Assoc Prf, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuce Y, Karakus SA, Simsek T, Onal C, Sezen O, Cevik B, Aydogmus E. Comparative efficacy of ultrasound-guided erector spinae plane block versus wound infiltration for postoperative analgesia in instrumented lumbar spinal surgeries. BMC Anesthesiol. 2024 Oct 15;24(1):374. doi: 10.1186/s12871-024-02754-9. PMID 39407122